CLINICAL TRIAL: NCT05323357
Title: Establishment of Human Organoid Lines as a Tool to Dissect Molecular Pathways of Host-microbiota Interactions
Brief Title: Bern Human Organoid-Study to Study Host-microbe Interaction
Acronym: humorg
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01865
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Organoids; Allergy and Immunology; Microbiota
Keywords: Enteroids; Host-Microbiota; Mucosal Immunology
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Biopsies from the Duodenum (routine Gastroscopy), Ileum (routine Colonoscopy) or Colon (routine Colonoscopy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The human body inhabits a complex consortium of different microbes which together form the microbiota. Virtually every surface of the human body is colonized by a distinct microbiota, forming complex communities. An increasing number of research results indicates that changes in the microbiota can have vast effects on the health of its host.

Most studies investigating the microbiota were conducted on animals, as many interventions and investigations cannot be performed on humans due to ethical considerations. This raises the question if findings from experimental studies are translational and can benefit patients. That becomes especially apparent when trying to dissect molecular mechanisms involved in this fine-tuned interplay between nutrients, the microbiota, and its host.

By establishing human organoid cultures from the large and small intestine that can be exposed to microbes and/or microbial products with subsequent transcriptomic, epigenetic and immunological analysis, the investigators aim to generate findings with high translational potential with new insights into the complex interaction of the microbiota, the host and its immune system.

DETAILED DESCRIPTION:
* Data obtained from participants will be recorded in the database Redcap to ensure high-quality data recording
* Establishment of human organoid cultures are standardized by published protocols (Pleguezuelos-Manzano et al. 2020)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Indication for upper or lower endoscopic procedure
* Ability to understand and follow study procedures and understand informed consent
* Age 18-80 years
* Negative pregnancy test result prior to study enrollment of female study participants (test will be performed prior to enrollment)
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Disease known to chronically affect gut microbiota, gut epithelium or gut-associated immune system, namely inflammatory bowel disease, diverticulitis, microscopic colitis, liver cirrhosis, malignancy within the digestive tract, systemic sclerosis, coeliac disease, common-variable immunodeficiency, diabetes mellitus
* Medication with immunosuppressants (e.g. corticoids, biological therapy)
* Current diagnosis of a hematological disorder (e.g. anemia with hemoglobin <7 g/dl, leukemia) or any other absolute contraindication for blood draw
* Women who are pregnant
* Serious coagulation disorder, relevant thrombocytopenia (<50'000/ul), double platelet-inhibition, oral anticoagulation (ASS therapy is possible)
* Known or suspected non-compliance, drug, or alcohol abuse
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons
* Inability or unwillingness to provide blood samples and tissue samples (biopsies)
* Participants taking oral anticoagulant or with bleeding disorders who would be at much higher risk of bleeding after biopsy samples or who are contraindicated for an endoscopic examination
* Patients unable to give informed consent
* Patients that have been under antibiotic therapy in the last 4 weeks
* Participation in other clinical study interfering with study procedures
* Potential study participants that wish not to be informed about random results acquired during the study (e.g., during endoscopy or genetic analysis) relevant for their health and for prevention of diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients undergoing routine ileo-colonoscopy without sign of inflammation, dysplasia, or neoplasia in histology
  2. Patients undergoing routine gastro-duodenoscopy without sign of inflammation, dysplasia, or neoplasia in histology
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in the transcriptomic profile of epithelial cells before and after organoid culture | 3 Years
  Assessment of changes in the transcriptomic profile of epithelial cells before and after organoid culture is established by RNA-sequencing and quantitative polymerase chain reaction (qPCR)
Assessment of changes in the epigenome of epithelial cells before and after organoid culture | 3 Years
  Assessment of changes in the epigenome of epithelial cells before and after organoid culture is established by whole genome bisulphite sequencing and chromatin immunoprecipitation sequencing
Transcriptomic and Epigenomic Landscape of host-microbiota Interaction | 3 Years
  Determining effects of microbial-derived metabolites on the transcriptomic and epigenomic landscape of human organoids treated with the respective metabolite
Host-Microbiota interaction - Stem cell maintenance and Cell Differentiation | 3 Years
  Determining effects of microbial-derived metabolites on epithelial cell differentiation and stem cell maintenance

SECONDARY OUTCOMES:
3D-to-2D Transwell System | 3 Years
  Establishing a method to transform human organoid culture into a 2-dimensional trans-well system which allows transportation studies, characterization of epithelial integrity and other downstream analysis
Gut-on-a-chip | 3 Years
  Applying 2-dimensional trans-well system to a gut-on-a-chip set-up in collaboration with the Artorg Center at the University of Bern

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ganal-Vonarburg, Prof, Principal Investigator — Inselspital, University Hospital Bern
Locations (1):
- Inselspital, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Pleguezuelos-Manzano C, Puschhof J, van den Brink S, Geurts V, Beumer J, Clevers H. Establishment and Culture of Human Intestinal Organoids Derived from Adult Stem Cells. Curr Protoc Immunol. 2020 Sep;130(1):e106. doi: 10.1002/cpim.106. PMID 32940424
- See also: Pleguezuelos-Manzano C et al. 2020 — https://pubmed.ncbi.nlm.nih.gov/32940424/